CLINICAL TRIAL: NCT00315601
Title: Comparison of the Intrapulmonary and Plasma Concentrations of Telithromycin and Azithromycin in Healthy Adult Subjects
Brief Title: Intrapulmonary Pharmacokinetics of Antibiotics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sanofi-Aventis wanted the study terminated.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Sanofi (Industry)
Responsible Party: University of Illinois at Chicago, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 2005-0748
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Telithromycin (drug); Azithromycin (drug); Bronchoalveolar lavage (procedure); Pharmacokinetics
MeSH Terms: interventions — telithromycin; Azithromycin; Bronchoalveolar Lavage; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Telithromycin — 800 mg once a day for 5 days
  Other Names: Ketek
Drug: azithromycin — 500 mg on day 1, and then 250 mg once-daily on days 2 through 5
  Other Names: Zithromax
Procedure: bronchoalveolar lavage — One bronchoscopy with bronchoalveolar lavage with each drug administration
  Other Names: Bronchoscopy with BAL
Drug: Telithromycin — Telithromycin 800 mg once a day
  Other Names: Ketek

SUMMARY:
The major objectives of this research are to see how much, and for how long, telithromycin and azithromycin get into the fluids and cells of the lung.

DETAILED DESCRIPTION:
The primary objective of this descriptive study is to determine and compare the plasma, epithelial lining fluid (ELF), and alveolar macrophage (AM) concentrations following multiple oral doses of telithromycin and azithromycin in healthy, non-smoking adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years, inclusive, of age
* No history of smoking within the last 1 year
* Body weight within +/- 15% of the Metropolitan Life Insurance Company tables
* No clinically important abnormalities in the medical history or physical exam
* Female subjects of childbearing potential must have a negative pregnancy test
* Female subjects of childbearing potential must use reliable methods of birth control

Exclusion Criteria:

* Allergy to telithromycin, azithromycin, or any macrolide antibiotic
* Allergy or serious adverse reactions to benzodiazepines or lidocaine
* History of renal, gastrointestinal, or liver disease
* Significant hypertension
* Clinically significant heart or pulmonary diseases
* History of drug or alcohol dependence within 12 months of study entry
* Positive pregnancy test
* Currently breast feeding
* Use of any drug within 2 weeks of study entry
* Received an investigational drug within 30 days of study entry

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Plasma and intrapulmonary drug concentrations and pharmacokinetic parameters | 7 days

SECONDARY OUTCOMES:
How long does the study antibiotics get into the fluids and cells of the lung. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Pharm.D., Principal Investigator — University of Illinois at Chicago; Mark H. Gotfried, M.D., Principal Investigator — Pulmonary Associates, PA; Larry H. Danziger, Pharm.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Pulmonary Associates PA, Phoenix, Arizona, United States